CLINICAL TRIAL: NCT06512935
Title: Ventilator Pressure and Optimization of Compliance and Hemodynamics: VPOCH Trial
Brief Title: Ventilator Pressure and Optimization of Compliance and Hemodynamics
Acronym: VPOCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kulsajan Singh Bhatia, Neonatal Perinatal Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300013132
Record Dates: First submitted 2024-07-05; First posted 2024-07-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Bronchopulmonary Dysplasia; Pulmonary Hypertension Due to Lung Diseases and Hypoxia; Extreme Prematurity; Ventilator Lung; Newborn; Ventilation Perfusion Mismatch
Keywords: Respiratory distress syndrome; ventilation mechanics in newborn; cardiac hemodynamics newborn
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Hypoxia; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Single centre, randomized crossover study. This study will include preterm infants with recovering RDS born at age < 34 weeks of gestational age on respiratory support via conventional mechanical ventilation or on HFJV.
  Infants will be randomized to the order of testing, increasing the PEEP (+1 cmH2O and +2 cmH2O) or decreasing the PEEP (+1 cmH2O and +2 cmH2O) with baseline measurements and Echo done at original PEEP and at each subsequent PEEP.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cardiac hemodynamics and respiratory status assessment with increasing PEEP (Experimental): Infants will be randomized to the order of changes in PEEP levels during mechanical ventilation - increase followed by decrease in PEEP.
  Baseline parameters looking into cardiac hemodynamics as well as compliance and respiratory mechanics will be assessed using EIT
  Interventions: Other: Increase in the PEEP followed by decrease in the PEEP
- cardiac hemodynamics and respiratory status assessment with decreasing PEEP (Active Comparator): Infants will be randomized to the order of changes in PEEP levels during mechanical ventilation - decrease followed by increase in PEEP.
  Baseline parameters looking into cardiac hemodynamics as well as compliance and respiratory mechanics will be assessed using EIT
  Interventions: Other: Decrease in the PEEP followed by increase in the PEEP

INTERVENTIONS:
Other: Increase in the PEEP followed by decrease in the PEEP — Changes in the ventilator PEEP and its effect on lung and cardiac hemodynamics
  Arms: cardiac hemodynamics and respiratory status assessment with increasing PEEP
Other: Decrease in the PEEP followed by increase in the PEEP — Changes in the ventilator PEEP and its effect on lung and cardiac hemodynamics
  Arms: cardiac hemodynamics and respiratory status assessment with decreasing PEEP

SUMMARY:
In preterm infants < 34 weeks' gestation at birth receiving respiratory support with invasive positive pressure ventilation, the positive end-expiratory pressure (PEEP) of best compliance will increase the cardiac output and improve oxygenation. This study may emphasize using point-of-care echocardiography along with electrical impedance tomography (EIT) to optimize ventilator settings in preterm infants.

Infants will be randomized to a 4-hour crossover period of increasing and decreasing PEEP in random order from baseline to determine compliance, oxygenation, and cardiac hemodynamics at each step using echocardiography (ECHO) and EIT measurements. There will be a 15-minute washout period after changes prior to data collection.

DETAILED DESCRIPTION:
In preterm infants < 34 weeks' gestation at birth receiving respiratory support with invasive positive pressure ventilation, the positive end-expiratory pressure (PEEP) of best compliance will increase the cardiac output and improve oxygenation. This study may emphasize using point-of-care echocardiography along with EIT to optimize ventilator settings in preterm infants.

Neonatal ventilation is a critical intervention to support breathing for newborns with respiratory distress syndrome (RDS), underdeveloped lungs, and evolving bronchopulmonary dysplasia (BPD). Positive airway pressure helps maintain patency of the airways and improves ventilation and oxygenation by maintaining the functional residual capacity (FRC) and keeping the alveoli patent. Peak inspiratory pressure (PIP) and positive end-expiratory pressure (PEEP) are terms commonly used in mechanical ventilation to describe the pressures applied to the respiratory system during the different phases of the breathing cycle. These parameters are essential in managing and optimizing ventilation for infants with respiratory failure.

This study will include preterm infants with recovering RDS born at age < 34 weeks of gestational age on respiratory support via conventional mechanical ventilation or on high-frequency jet ventilation (HFJV). Infants will be randomized to the order of testing, increasing the PEEP (+1 cmH2O and +2 cmH2O) or decreasing the PEEP (+1 cmH2O and +2 cmH2O) with baseline measurements and Echo done at original PEEP and each subsequent PEEP.

Following informed consent, randomization will be performed using sequentially numbered sealed opaque envelopes. The randomization envelope will be signed before it is opened just before starting the study on each infant to indicate the first intervention for the infant.

This will be a single-center, randomized crossover study. The randomization envelope will be signed before it is opened just before starting the study on each infant to indicate the first intervention for the infant.

Randomization will occur after a baseline assessment of cardiac hemodynamics and respiratory status at the current set PEEP level. Infants will be randomized to the order of changes in PEEP levels during mechanical ventilation - increase followed by decrease versus decrease followed by increase. Randomization will use opaque sealed envelopes of varying block sizes from 2-4 with a 1:1:1:1 allocation ratio.

Infants will be randomized to a 4-hour crossover period of increasing and decreasing PEEP in random order from baseline and there will be a 15-minute washout period after changes before data collection.

All infants enrolled in the study will have routine monitoring, uniform target saturation ranges of 91-95% with alarm limits set at 88-95%, and standard care for the duration of the study. Pulse oximetry recordings will be downloaded using ixTrend (iexcellence, Wildau, Germany) software to a secure computer system for later data analysis.

Infants will continue standard treatment as recommended by the treating physician and will act as their own controls.

Primary secondary outcomes are described below. Electrical impedance tomography data will be collected in the Syntec machine and safely secured in the university computer system. Pulse oximetry recordings will be downloaded using ixTrend software to a secure computer system for later data analysis.

ECHO results will be stored in the unit ECHO machine and results will be reported by certified cardiologists blinded to the data collected to improve the study design's internal and external validity.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants with recovering respiratory distress syndrome (RDS) who were born at a gestational age < 34 weeks and are receiving respiratory support via conventional mechanical ventilation or on HFJV.

* Post-natal age > 7 days and less than 1 month (outside golden week protocol)
* Gestational age ≥ 21 weeks and ≤ 34 week
* Infants with written informed consent obtained from legal guardian

Exclusion Criteria:

* Blood culture-positive sepsis
* Congenital anomalies affecting respiration
* Cyanotic or ductal-dependent congenital heart disease
* Newborns who are considered too unstable for study enrolment per neonatology attending
* Newborns on pressors or steroids for maintaining cardiac output
* Non-invasive ventilation or newborn with significant BPD (bronchopulmonary dysplasia) with pulmonary hypertension (HTN)
* Open skin wounds or abrasions on the chest wall.

Ages: 7 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac index with increase/decrease in PEEP as measured by ECHO and EIT | During a 4 hour cross-over period on either intervention
PEEP of best compliance and best oxygenation as per EIT measurements | During a 4 hour cross-over period on either intervention

SECONDARY OUTCOMES:
Tidal volume variation | During a 4 hour cross-over period on either intervention
Oxygen saturation index | During a 4 hour cross-over period on either intervention
End-expiratory lung impedance (EELI), End-inspiratory lung impedance (EILI) | During a 4 hour cross-over period on either intervention
Transcutaneous carbon dioxide (TcCO2) values in response to varying PEEP levels | During a 4 hour cross-over period on either intervention
Respiratory Severity Score (RSS) | During a 4 hour cross-over period on either intervention
  RSS: mean airway pressure (MAP) x fraction of inspired oxygen (FiO2)
oxygen saturation (SpO2) values | During a 4 hour cross-over period on either intervention
% tidal distribution | During a 4 hour cross-over period on either intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kulsajan S Bhatia, MD, Principal Investigator — University of Alabama at Birmingham; Colm P Travers, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Univerisity of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No